CLINICAL TRIAL: NCT06690112
Title: A Pilot Study Comparing the Incidence of Intra-abdominal Complications According to the Removal of the Drainage Tube in Patients With Large Amounts of Drainage After Gastrectomy in Gastric Cancer Patients
Brief Title: Pilot Study for High Output Drainage Removal After Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2023-0393
Record Dates: First submitted 2024-10-29; First posted 2024-11-15 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
Keywords: Drainage tube; Gastrectomy; High output
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drainage removal group (Experimental): Patients who remove their draiange tube at discharge
  Interventions: Procedure: Arm I (Drainage tube removal)
- Drainage maintain group (No Intervention): Patients who maintain their draiange tube at discharge

INTERVENTIONS:
Procedure: Arm I (Drainage tube removal) — During gastrectomy, a drainage tube is placed within the abdominal cavity. In Arm I (the intervention group), the drainage tube will be removed at the bedside. This procedure is a simple intervention that does not require local anesthesia and involves the removal of the drainage tube by cutting the nylon suture.
  Arms: Drainage removal group

SUMMARY:
*Objective: The study aims to evaluate whether there is a difference in intra-abdominal complication rates between patients discharged with or without a drainage tube following gastrectomy with high postoperative drainage (≥300ml/day).

*Study Design: This is an open-label randomized controlled trial (RCT) involving two groups. Patients will be randomly assigned to either maintain the drainage tube (control) or have it removed (experimental) before discharge. The primary endpoint is the incidence of intra-abdominal complications within one month post-surgery.

*Participants:

The study targets 60 patients (30 per group) who meet the following criteria:

Diagnosed with gastric adenocarcinoma and underwent curative gastrectomy (R0 resection).

Postoperative drainage of 300-500 ml/day on the 4th day after surgery. Patients with stage IV cancer, peritoneal metastasis, or postoperative complications requiring additional intervention are excluded.

*Methods: All participants will follow standard postoperative care except for the removal or retention of the drainage tube. Follow-up will occur at 1 and 3 weeks post-discharge, with clinical examinations and imaging (if necessary) to monitor for complications such as infection or abscess. The study's total observation period will last four weeks from the surgery date.

*Data Collection: Data will include patient demographics, surgical details, postoperative management, and the occurrence of complications. Drainage volumes will be recorded daily for those discharged with a tube, and tube removal will occur based on specific criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients pathologically diagnosed with gastric adenocarcinoma before surgery.
* Patients eligible for complete surgical resection (R0 resection).
* Patients with an ASA (American Society of Anesthesiologists) score of 3 or lower.
* Patients with more than 300 ml of drainage in the 24 hours on the postoperative day 4.

Exclusion Criteria:

* Patients aged 80 or older.
* Patients with stage IV gastric cancer.
* Patients with ascites due to peritoneal metastasis.
* Patients with evident intra-abdominal complications following surgery.
* Patients who require the insertion of additional percutaneous drainage due to insufficient drainage.
* Patients who underwent incomplete gastric resection (R1 or R2 resection).
* Patients diagnosed with cancers other than gastric cancer.
* Patients with a history of major intra-abdominal surgery or abdominal radiotherapy that may hinder the normal absorption of intra-abdominal fluid.
* Patients with more than 500 ml of drainage in the 24 hours on postoperative day 4.
* Patients presenting with any of the following clinical signs or diagnoses:

  1. Postoperative pancreatic fistula (POPF), defined as drain amylase levels (Drain amylase; D-amy) more than 3 times higher than serum amylase levels (Serum amylase; S-amy).
  2. Fever exceeding 37.8℃.
  3. Presence of any of the following clinical markers of inflammation:

     i. White blood cell count (WBC) > 15,000/μL ii. C-reactive protein > 200 mg/L
  4. Observation of non-serous drainage fluid, such as:

     i. Chylous fluid: Milky-colored fluid. ii. Bloody or sanguineous fluid: Intra-abdominal fluid suggestive of ongoing hemorrhage.
* Vulnerable subjects will not be enrolled in the study, including minors, pregnant women, neonates, adults with impaired consent capacity, individuals in institutional facilities, students, employees of medical institutions or research centers, pharmaceutical company employees, military personnel, unemployed persons, impoverished individuals, homeless individuals, terminally ill patients, or patients in emergency situations.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intra-Abdominal Complications | up to 1 month
  Complications include infections, abscesses, or any clinically significant intra-abdominal issues that require medical intervention.

SECONDARY OUTCOMES:
Drain-Related Complications | up to 1month
  The occurrence of complications related to the drainage tube in the control group, such as infection at the insertion site or mechanical issues.
CRP Level Changes | up to 1month
  The comparison of C-reactive protein (CRP) level changes between the intervention and control groups during the 4-week postoperative follow-up. CRP levels will be measured to assess inflammation and potential early signs of complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severacne Hospital Yonsei University College of Medicine, Seoul, South Korea